CLINICAL TRIAL: NCT04115527
Title: A Prospective Randomized Controlled Study Comparing Standard and Extended Lymphadenectomy for Pancreatic Head Cancer
Brief Title: Should a Standard Lymphadenectomy Include the No. 16 Lymph Nodes for Patients With Pancreatic Head Adenocarcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weishen WANG, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBP-RCT-003
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: RCT; Standard lymphadenectomy; Extended lymphadenectomy; Pancreaticoduodenectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard lymphadenectomy (Active Comparator): Standard lymphadenectomy includes No 5 6 8a 12b1 12b2 12c 13a 13b 14a 14b 17a 17b lymph nodes harvested during the pancreaticoduodenectomy with CHILD's digestive reconstruction
  Interventions: Procedure: Standard Lymphadenectomy
- Extended lymphadenectomy (Experimental): In addition to the standard lymphadenectomy, para-aortic lymph nodes (No16) is included, in particular No 16b1 lymph nodes (Lymph nodes along the psterior side of the pancreas between the aorta and inferior vena cava).
  Interventions: Procedure: Extended Lymphadenectomy

INTERVENTIONS:
Procedure: Extended Lymphadenectomy — Lymph node dissection includes No 5 6 8a 12b1 12b2 12c 13a 13b 14a 14b 16 17a 17b lymph nodes
  Arms: Extended lymphadenectomy
Procedure: Standard Lymphadenectomy — Lymph node dissection includes No 5 6 8a 12b1 12b2 12c 13a 13b 14a 14b 17a 17b lymph nodes
  Arms: Standard lymphadenectomy

SUMMARY:
The aim of this study is to determine whether para-aortic lymph nodes(No.16) should be included in the lymphadenectomy during the pancreatoduodenectomy in order to improve the long-term survival of patients with pancreatic head ductal adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic cancer is now raised to the 7th leading cause of death. Surgical resection seems to be the unique curative therapy for pancreatic cancer. The pancreaticoduodenectomy is widely performed for the patients with pancreatic head cancer in recent decades. The lymphadenectomy is an indispensible procedure. In 2014, the International Study Group for Pancreatic Surgery (ISGPS) recommended a standard lymphadenectomy should include lymph node stations 5, 6, 8a, 12b1, 12b2, 12c, 13a, 13b, 14a, 14b, 17a, and 17b. However, no consensus was reached on Lymph node 16 in particular 16b1. There was no stronge evidence available concerning the impact on survival.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of pancreatic ductal adenocarcinoma
* Signed the informed consents

Exclusion Criteria:

* Pathologic diagnosis of other pancreatic cancers
* Pre-operative anti-cancer treatment
* Recurrence patients
* Patients with contraindication(hepatic/ respiratory/ renal dysfunction, etc )
* Pre operative exam: Total bilirubin more than 250µmol/L
* AJCC stage IV
* Operation non radical

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year overall survival rate | 1 year post-operation
  1 year overall survival rate
3 years overall survival rate | 3 years post-operation
  3 years overall survival rate
5 years overall survival rate | 5 years post-operation
  5 years overall survival rate

SECONDARY OUTCOMES:
Postoperative Complications | Within 90 days or before discharge
  pancreatic fistula, bile leakage, haemorrhage, DGE, etc
1, 3 & 5 years disease free survival rate | 1, 3 & 5 years post-operation
  1, 3 & 5 years disease free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Jiancheng WANG, Dr, Study Director — Shanghai Ruijin Pancreatic Disease Center
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided